CLINICAL TRIAL: NCT02016716
Title: A Multicenter, Randomized, Multiple-dose Phase 3 Study to Evaluate the Noninferiority of Romosozumab at a 90 mg/mL Concentration Compared With a 70 mg/mL Concentration in Postmenopausal Women With Osteoporosis
Brief Title: A Randomized Phase 3 Study to Evaluate Two Formulations of Romosozumab in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20120156; 2013-000434-35 (EudraCT Number)
Record Dates: First submitted 2013-12-10; First posted 2013-12-20 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-09

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Romosozumab 90 mg/mL (Experimental): Participants received 210 mg romosozumab monthly, administered as 2 subcutaneous (SC) 1.17 mL injections of a 90 mg/mL solution, for 6 months.
  Interventions: Drug: Romosozumab 90 mg/mL
- Placebo 90 mg/mL (Experimental): Participants received matching placebo administered as 2 subcutaneous injections of 1.17 mL every month for 6 months.
  Interventions: Drug: Placebo 90 mg/mL
- Romosozumab 70 mg/mL (Experimental): Participants received 210 mg romosozumab monthly, administered as 3 subcutaneous 1.0 mL injections of a 70 mg/mL solution, for 6 months.
  Interventions: Drug: Romosozumab 70 mg/mL
- Placebo 70 mg/mL (Placebo Comparator): Participants received matching placebo administered as 3 subcutaneous injections of 1.0 mL every month for 6 months.
  Interventions: Drug: Placebo 70 mg/mL

INTERVENTIONS:
Drug: Romosozumab 90 mg/mL — Administered as 2 SC injections of a 90 mg/mL concentration in a 1.17 mL crystal zenith resin prefilled syringe (PFS).
  Other Names: AMG 785; EVENITY™
  Arms: Romosozumab 90 mg/mL
Drug: Placebo 90 mg/mL — Placebo administered as 2 SC injections with the 1.17 mL crystal zenith resin PFS.
  Arms: Placebo 90 mg/mL
Drug: Romosozumab 70 mg/mL — Administered as 3 SC injections of a 70 mg/mL concentration in a 1.0 mL glass PFS.
  Other Names: AMG 785; EVENITY™
  Arms: Romosozumab 70 mg/mL
Drug: Placebo 70 mg/mL — Placebo administered as 3 SC injections with the 1.0 mL glass PFS.
  Arms: Placebo 70 mg/mL

SUMMARY:
The purpose of this study is to compare 2 formulations of romosozumab (AMG 785) on bone mineral density (BMD) in postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
Upon confirmation of eligibility, participants were randomized in a 22:5:22:5 ratio to the following treatment groups:

* Romosozumab 90 mg/mL
* Placebo 90 mg/mL
* Romosozumab 70 mg/mL
* Placebo 70 mg/mL

After completing a 6-month treatment period, participants entered a 3-month follow-up period with an end of study (EOS) at month 9.

For the analysis of efficacy endpoints, the 2 placebo groups were combined into a single placebo group. For safety analyses, the data for placebo were presented separately for each group.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women with osteoporosis at high risk for fracture defined as

* BMD T-score ≤ -2.50 at the lumbar spine, total hip, or femoral neck AND
* a history of fragility fracture or at least 2 other risk factors

Exclusion Criteria:

* BMD T score < -3.50 at the total hip or femoral neck.
* History of hip fracture.
* History of metabolic or bone disease (except osteoporosis).
* Use of agents affecting bone metabolism.
* Vitamin D insufficiency.
* History of solid organ or bone marrow transplants.
* Hyper- or hypocalcemia.
* Hyper- or hypothyroidism.
* Hyper- or hypoparathyroidism.

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2014-09-08 (Actual); Study Completion 2014-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- United States (2):
  - Research Site, Gainesville, Georgia
  - Research Site, Bethesda, Maryland
- Czechia (3):
  - Research Site, Brno
  - Research Site, Klatovy
  - Research Site, Uherské Hradiště
- Poland (7):
  - Research Site, Gdynia
  - Research Site, Gliwice
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Świdnik
  - Research Site, Warsaw
  - Research Site, Wroclaw

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 centers: 7 in Poland, 2 in the Czech Republic, and 2 in the United States. The first participant enrolled on 03 December 2013 and the last participant enrolled on 07 March 2014.
Pre-assignment Details: Eligible participants were randomized in a 22:5:22:5 ratio to receive
  * romosozumab 90 mg/mL
  * placebo 90 mg/mL
  * romosozumab 70 mg/mL
  * placebo 70 mg/mL
  For efficacy analyses the 2 placebo groups were combined, for safety analyses the data were reported separately.
Groups:
- Placebo: Participants received matching placebo (either administered as 2 subcutaneous (SC) injections of 1.17 mL or 3 SC injections of 1.0 mL) every month for 6 months.
- Romosozumab 70 mg/mL: Participants received 210 mg romosozumab monthly, administered as 3 subcutaneous 1 mL injections of a 70 mg/mL solution, for 6 months.
- Romosozumab 90 mg/mL: Participants received 210 mg romosozumab monthly, administered as 2 subcutaneous 1.17 mL injections of a 90 mg/mL solution, for 6 months.
Period: Overall Study
Arm/Group | Placebo | Romosozumab 70 mg/mL | Romosozumab 90 mg/mL
Started | 53 | 118 | 123
Received Study Treatment | 53 | 118 | 123
Completed | 47 | 110 | 117
Not Completed | 6 | 8 | 6
Not completed — Withdrawal by Subject | 5 | 5 | 5
Not completed — Protocol-specified Criteria | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants (full analysis set)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romosozumab 70 mg/mL | Romosozumab 90 mg/mL | Total
Number analyzed (Participants) | 53 | 118 | 123 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.0) | 67.4 (7.1) | 67.7 (7.6) | 67.7 (7.5)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 23 | 46 | 46 | 115
  ≥ 65 years | 30 | 72 | 77 | 179
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 118 | 123 | 294
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 9 | 17
  Not Hispanic or Latino | 51 | 112 | 114 | 277
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 2 | 0 | 2
  Black (or African American) | 0 | 1 | 0 | 1
  White | 53 | 115 | 123 | 291
Lumbar Spine Bone Mineral Density (BMD) T-score [Mean (Standard Deviation); unit: T-score] — The T-score is the bone mineral density (BMD) at the site when compared to that of a healthy thirty-year-old. Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman.
  T-score | -2.842 (1.033) | -2.965 (0.960) | -3.029 (0.687) | -2.970 (0.871)
Total Hip BMD T-score [Mean (Standard Deviation); unit: T-score] | -2.057 (0.634) | -1.819 (0.673) | -1.828 (0.649) | -1.866 (0.660)
Femoral Neck BMD T-score [Mean (Standard Deviation); unit: T-score] | -2.304 (0.517) | -2.139 (0.611) | -2.018 (0.593) | -2.118 (0.595)
Serum Procollagen Type 1 N-telopeptide (P1NP) [Median (Inter-Quartile Range); unit: μg/L] — Population: Participants with available data
  μg/L
    number analyzed (Participants) | 53 | 117 | 123 | 293
    (all) | 49.0 [38.0 to 61.0] | 53.0 [40.0 to 61.0] | 50.0 [40.0 to 64.0] | 51.0 [40.0 to 63.0]
Serum Type 1 Collagen C-telopeptide (CTX) [Median (Inter-Quartile Range); unit: ng/L] — Population: Participants with available data
  ng/L
    number analyzed (Participants) | 52 | 117 | 123 | 292
    (all) | 426.5 [296.5 to 560.5] | 440.0 [288.0 to 613.0] | 402.0 [299.0 to 530.0] | 426.0 [295.0 to 590.0]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) at the Lumbar Spine
Description: Bone mineral density was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and month 6
Population: All randomized participants who had a baseline and a month 6 lumbar spine DXA BMD measurement
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg/mL | Romosozumab 90 mg/mL
Number analyzed (Participants) | 46 | 110 | 117
percent change | 0.8 [-0.4 to 2.1] | 9.6 [8.8 to 10.4] | 9.2 [8.4 to 10.0]
Statistical Analysis 1: Comparison: Romosozumab 70 mg/mL vs Romosozumab 90 mg/mL; The primary hypothesis was that the mean percent change from baseline in lumbar spine BMD at month 6 in participants receiving romosozumab 210 mg QM using the 90 mg/mL concentration would not be inferior to that in participants receiving romosozumab 210 mg QM using the 70 mg/mL concentration; Test type: Non-Inferiority — Non-inferiority was claimed if the lower bound of the 1-sided 97.5% CI (or the lower bound of 2-sided 95% CI) of the mean difference between the 2 romosozumab groups was > -2.0%; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-1.5 to 0.7] — Based on ANCOVA model adjusting for treatment, and baseline lumbar spine BMD T-score

2. Secondary Outcome: Percent Change From Baseline in Total Hip BMD
Description: Total hip BMD was measured using DXA. The analysis was based on an ANCOVA model adjusted for treatment and baseline total hip BMD T-score.
Time Frame: Baseline and month 6
Population: All randomized participants who had a baseline and month 6 hip DXA BMD measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg/mL | Romosozumab 90 mg/mL
Number analyzed (Participants) | 46 | 110 | 116
percent change | -0.0 [-0.9 to 0.8] | 3.9 [3.4 to 4.4] | 3.4 [2.9 to 4.0]

3. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD
Description: Femoral neck BMD was measured using DXA. The analysis was based on an ANCOVA model adjusted for treatment and baseline femoral neck BMD T-score.
Time Frame: Baseline and month 6
Population: All randomized participants who had a baseline and month 6 femoral neck DXA BMD measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg/mL | Romosozumab 90 mg/mL
Number analyzed (Participants) | 46 | 110 | 116
percent change | -0.5 [-1.5 to 0.5] | 3.1 [2.5 to 3.8] | 2.6 [2.0 to 3.3]

4. Secondary Outcome: Percent Change From Baseline in N-Terminal Propeptide Type 1 Procollagen (P1NP)
Time Frame: Baseline, month 1, month 3, and month 6
Population: All randomized participants who had a baseline and at least one postbaseline measurement for P1NP, and with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg/mL | Romosozumab 90 mg/mL
Number analyzed (Participants) | 51 | 115 | 120
percent change
  Month 1: number analyzed (Participants) | 51 | 111 | 116
  Month 1 | 2.000 [-5.797 to 16.129] | 96.296 [67.143 to 159.341] | 97.435 [69.259 to 126.179]
  Month 3: number analyzed (Participants) | 48 | 110 | 115
  Month 3 | -9.601 [-21.503 to 2.922] | 23.960 [-1.587 to 46.667] | 16.216 [-10.390 to 50.000]
  Month 6: number analyzed (Participants) | 45 | 102 | 110
  Month 6 | -12.500 [-27.500 to 14.286] | -2.885 [-28.070 to 18.421] | -3.604 [-22.222 to 27.273]

5. Secondary Outcome: Percent Change From Baseline in Serum C-Telopeptide (CTX)
Time Frame: Baseline, month 1, month 3, and month 6
Population: All randomized participants who had a baseline and at least one postbaseline measurement for CTX and with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg/mL | Romosozumab 90 mg/mL
Number analyzed (Participants) | 51 | 115 | 120
percent change
  Month 1: number analyzed (Participants) | 51 | 111 | 117
  Month 1 | 0.282 [-16.183 to 12.874] | -23.158 [-42.943 to -9.967] | -21.456 [-35.602 to -7.246]
  Month 3: number analyzed (Participants) | 48 | 110 | 116
  Month 3 | -5.687 [-20.666 to 15.566] | -11.219 [-35.206 to 9.484] | -5.473 [-24.139 to 26.386]
  Month 6: number analyzed (Participants) | 45 | 108 | 114
  Month 6 | -8.120 [-26.935 to 10.059] | -25.780 [-43.573 to -8.216] | -17.305 [-37.566 to 6.405]

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the first dose of study drug until 90 days after last dose (9 months overall).
Description: One participant was randomized to the placebo group but incorrectly received 1 dose of romosozumab 70 mg/mL and was included in the romosozumab 70 mg/mL group for analysis of adverse events.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Placebo 70 mg: Participants received matching placebo administered as 3 subcutaneous injections of 1.0 mL every month for 6 months.
Arm/Group | Placebo 70 mg | Placebo 90 mg/mL | Romosozumab 70 mg/mL | Romosozumab 90 mg/mL
Serious Adverse Events (participants affected / at risk) | 4/26 | 2/26 | 7/119 | 3/123
Other Adverse Events (participants affected / at risk) | 9/26 | 5/26 | 24/119 | 38/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 70 mg (N=26) | Placebo 90 mg/mL (N=26) | Romosozumab 70 mg/mL (N=119) | Romosozumab 90 mg/mL (N=123)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Appendicitis noninfective (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mesenteric artery embolism (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Retrograde amnesia (Nervous system disorders) | 1 | 0 | 0 | 0
Umbilical hernia repair (Surgical and medical procedures) | 0 | 0 | 1 | 0
Arterial rupture (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 70 mg (N=26) | Placebo 90 mg/mL (N=26) | Romosozumab 70 mg/mL (N=119) | Romosozumab 90 mg/mL (N=123)
Asthenia (General disorders) | 0 | 2 | 4 | 4
Injection site erythema (General disorders) | 0 | 0 | 2 | 7
Injection site pain (General disorders) | 0 | 0 | 7 | 3
Nasopharyngitis (Infections and infestations) | 3 | 0 | 9 | 19
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 7
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 2
Headache (Nervous system disorders) | 3 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.